CLINICAL TRIAL: NCT05230043
Title: The Choice of a Violent Suicidal Means: a MRI Study With Computational Modeling of Decision-making
Acronym: SUICIDE_DECIDE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2020/FJ-001; 2020-A03353-36 (Other: ANSM)
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Suicide, Attempted
Keywords: Neuroimaging; decision-making
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and hair samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Suicide Attempters using Violent Means: A violent suicidal act is any suicidal act conducted with any means except for medication overdose or superficial wrist cutting.
  Interventions: Other: Algometer test; Other: functional MRI
- Patient Control
  Interventions: Other: Algometer test; Other: functional MRI
- Healthy Controls
  Interventions: Other: Algometer test; Other: functional MRI
- Suicide Attempters not using Violent Means
  Interventions: Other: Algometer test; Other: functional MRI

INTERVENTIONS:
Other: Algometer test — The computerized pressure algometer, AlgoMed (Medoc, Ramat Yishai, Israel), will be used for mechanical pain stimulation to assess information about pain threshold and tolerance. A constant rate of pressure is delivered by the examiner, and the pressure is recorded in Kilopascal (kPa). The stimulation will be applied between the medial and distal joints of the phalanges of the dominant hand.
Other: functional MRI — * Two 8s sequences of spin echo field map with phase encoding AP and PA
  * A 12:00min bold sequence for resting-state
  * A 15:12min bold sequence for gambling task thickness=2mm, Matrix Size = 105×105, FOV=210×210mm2;
  * A 6:38min T1w MPR sequence
  * A 7:40min T1w MPR sequence
  * A 5:57min T2w SPC sequence
  * A 8:24min T2w SPC sequence
  * A 8:32min FLAIR T2w sequence
  * Two 8:26min Multi-echo GRE sequence
  * A 8:29min high resolution multi-echo GRE sequence
  * Two 6:46min multi-echo GRE sequence with and without magnetic transfer contrast
  * Two 6:03min diffusion weighted images with phase encoding AP and PA

SUMMARY:
The study authors hypothesize a combination of cognitive, brain structural, brain functional and brain connectivity impairments in Suicide Attempters compared to Patient Controls and Healthy Controls, with deficits more marked in suicide attempters using violent suicidal means including:

1. Impaired choices at the reversal learning task with responses influenced by immediate outcome. This deficit would be correlated with brain activity in ventromedial Prefrontal Cortex during resting state and with several peripheral markers of the 5HT-system.
2. Reduced loss aversion. These deficits would be related to altered dynamics of Blood-Oxygen Level Dependent signal in the dorsal and ventral striatum as well as in ventral Prefrontal Cortex/ orbitofrontal cortex during the loss aversion task. These deficits would also be correlated with several peripheral markers of the 5HT-system.
3. Increased pain tolerance facilitating the execution of a violent and possibly painful act. These deficits measured with the algometer would be correlated with several peripheral markers of the 5HT-system.
4. Reduced behavioral inhibition in aversive context at the orthogonalized GoNoGo task facilitating the choice of a violent means. These deficits would be associated with altered Blood-Oxygen Level Dependent signal in ventral Prefrontal Cortex/ orbitofrontal cortex and parietal cortex during the resting state and correlated with several peripheral markers of the 5HT-system.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (as assessed with the Edinburgh Handedness Scale).
* Agreement to participate and sign the informed consent form.
* Is insured or beneficiary of a health insurance plan.
* Speaks French.
* Suicide Attempters using Violent Means group:

  * a personal history of mood disorder (bipolar disorder or depressive disorders according to DSM-5 criteria measured with the MINI 7.0);
  * at least one suicidal act committed with a violent means within the last 5 years.
* Suicide Attempters using Non-Violent Means group:

  * a personal history of mood disorder (bipolar disorder or depressive disorders according to DSM-5 criteria measured with the MINI 7.0);
  * at least one suicidal act conducted within the last 5 years;
  * no lifetime history of suicidal act with a violent means.
* Patient Control group:

  * a personal history of mood disorder (bipolar disorder or depressive disorders according to DSM-5 criteria measured with the MINI 7.0);
  * never attempted suicide in their lifetime;
  * no family history of suicidal behavior up to the second biological degree.
* Healthy Control group:

  * no personal history of major mental disorder according to the MINI 7.0;
  * never attempted suicide in their lifetime;
  * no family history of suicidal behavior up to the second biological degree.

Exclusion Criteria:

* Current participation or in the exclusion period of another research protocol in a category 1 RIPH
* Currently under judicial protection, or under adult guardianship.
* Refusal to participate.
* Is pregnant or breast feeding.
* The suicide attempt may have impacted the brain functioning (e.g. following hanging, asphyxia by drowning, head trauma following jumping from height, bullet impact, etc). This criteria will be assessed clinically by the investigator.
* Mental retardation (known or observed during the interview).
* Current psychotic disorder (according to the MINI 7.0).
* Current hypomanic episode (according to the MINI 7.0).
* Current manic, mixed, rapid cycling episodes (according to the MINI 7.0).
* Alcohol or substance disorder within last 3 months (according to the MINI 7.0).
* Past major brain trauma (with loss of consciousness > 1 minute).
* Contra-indication to MRI (metal in body (including due to suicidal act), claustrophobia, impossibility to lie still on the back during one hour).
* Electroconvulsive therapy within the last three months.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Four groups of participants will be recruited:
  1. 20 individuals with personal history of mood disorder (bipolar disorder or depressive disorders) and at least one suicidal act committed with a violent means within the last 12 months.
  2. 20 individuals with personal history of mood disorder (bipolar disorder or depressive disorders) and at least one suicidal act conducted within the last 12 months but no lifetime history of suicidal act with a violent means.
  3. 20 individuals with personal history of mood disorder (bipolar disorder or depressive disorders) who never attempted suicide and have no family history of suicidal behavior up to the second biological degree.
  4. 20 individuals with no personal history of major mental disorder or suicidal act and no family history of suicidal behavior up to the second biological degree.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Brain activity between groups | Day 0
  Magnetic Resonance Imaging signal during the resting state and loss aversion task Blood-Oxygen Level Dependent sequences.

SECONDARY OUTCOMES:
Impaired reversal learning between groups | Day 0
  Proportion of participants in each group reaching the learning criterion of the Reversal learning task (8 consecutive correct trials) in each stage (acquisition and reversal).
Loss aversion between groups | Day 1
  Level of acceptance/reject rate according to the size of the potential gain and loss in each trial of the Loss aversion task
Pain tolerance between groups | Day 0
  Pressure pain tolerance threshold (mean of 3 consecutive trials) measured by algometer
Behavioral inhibition in aversive context between groups | Day 0
  Response latencies in the reward-only condition vs. the reward+punishment condition in the inforced categorization task

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jollant, Study Director — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Result] Jollant F, Leon C. Suicidal transition rates and their predictors in the adult general population: a repeated survey over 21 years in France. Eur Psychiatry. 2024 Oct 29;67(1):e74. doi: 10.1192/j.eurpsy.2024.1782. PMID 39468715